CLINICAL TRIAL: NCT06075381
Title: Safety and Efficacy of the Pulmonary Expansion Device (PED): A Novel Postoperative Pulmonary Reexpansion Strategy Using Negative Pressure Generation for the Management of Tracheostomized Patients - Phase 2 Study
Brief Title: Pulmonary Expansion Device in Tracheostomized Patients Therapies in Tracheostomized Patients
Acronym: PEDTRAQ
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02129
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Complications; Rehabilitation; Postoperative Care
Keywords: Inspiratory Capacity; Breathing Exercises; Self-help Devices; Inventions
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Controlled, randomized, blinded, parallel-group, Phase II clinical study of applying conventional management plus the use of a lung reexpansion device versus conventional management alone as a lung reexpansion strategy in tracheostomized patients.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not feasible to mask the treatment in the control group and intervention group, although both groups will receive a standard treatment. One group will receive treatment through the use of the PED, while the other group will receive treatment through intermittent positive pressure in cases of lung atelectasis or mild persistent hypoxemia.
  After obtaining informed consent from eligible participants, the assignment to the therapeutic group will be carried out using a code that does not openly indicate the assigned group. Individuals aware of the assignment will be the physiotherapists administering the interventions and collecting data in the electronic format, which will be isolated from the data analysis. Generating these codes for each patient aims to blind the interventions during the statistical analysis process. All information will be recorded in electronic format.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional management plus Pulmonary Expansion Device (PED) (Experimental): The conventional management used in the intensive care unit as a lung expansion strategy in patients with tracheostomy plus Pulmonary Expansion Device (PED).
  Interventions: Combination Product: Pulmonary Expansion Device (PED); Procedure: Conventional management
- Conventional management alone (Active Comparator): Conventional management employed in the intensive care unit as a lung expansion strategy in tracheostomized patients, without utilizing the Pulmonary Expansion Device (PED).
  Interventions: Procedure: Conventional management

INTERVENTIONS:
Combination Product: Pulmonary Expansion Device (PED) — The Pulmonary Expansion Device constitutes an innovative instrumental technique for lung expansion, designed for use in patients with or without an artificial airway. This device is attached to the artificial airway, the oronasal mask, or the patient's mouth. It enables voluntary control through a system of one-way valves that restrict the air's escape from the lungs to the outside. This creates an environment conducive to retaining air within the lungs, thereby increasing intrapulmonary pressure. Additionally, it reduces the risk of pulmonary complications associated with conventional management, employing a strategy free from exogenous application of positive pressure to the airway. This approach doesn't necessitate expensive equipment or electrical power.
  Arms: Conventional management plus Pulmonary Expansion Device (PED)
Procedure: Conventional management — The conventional management includes: Adequate postoperative pain control, global postural reeducation, reeducation of breathing pattern, airway hygiene, early mobilization, respiratory and scapular waist exercises, and in patients with evidence of lung atelectasis or mild persistent hypoxemia, conventional management will involve the use of intermittent positive pressure ventilation in the airway.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of using PED (Pulmonary Expansion Device) in tracheostomized patients requiring lung reexpansion therapy within a single institution. The main question it aims to answer is: In tracheostomized patients requiring lung reexpansion therapy, does the utilization of PED (Pulmonary Expansion Device) alongside conventional management constitute a safe and effective strategy for improving oxygenation, lung volumes, and reducing postoperative pulmonary complications, as compared to traditional management alone?

Researchers will compare lung expansion therapy with PED plus conventional management versus lung expansion therapy through conventional management in tracheostomized patients to assess the safety and efficacy in terms of improvement in oxygenation, lung volumes, and reduction of postoperative pulmonary complications.

DETAILED DESCRIPTION:
Sample size: Considering that the utilization of the PED introduces an innovative approach to the standard postoperative care of tracheostomized patients, who inherently face an elevated risk of pulmonary complications due to glottis derivation and are unable to engage in traditional respiratory exercises, there is currently an absence of information within the reviewed scientific literature concerning any device employed for evaluating gasometry and lung volume within this specific target population. Consequently, a comparable population that has undergone lung reexpansion techniques is not present for reference in this context. Therefore, when it comes to calculating the sample size, our only available reference is our pilot study involving 10 tracheostomized patients who underwent a lung reexpansion strategy using the PED. This study demonstrated noticeable improvements in oxygenation and lung volumes without encountering any related complications.

As a result, the sample size for this feasibility study has been adjusted based on the number of recently tracheostomized patients admitted to the Adult Intensive Care Unit. Concurrently in the immediate postoperative phase following thoracic surgery (41 patients) or high abdominal surgery (16 patients) throughout the year 2021. Consequently, it was determined that data would be collected from a cohort of 50 patients who meet the predefined inclusion criteria over one year. Both the intervention and control groups will be randomized equally. This Phase 2 study aims to provide essential feasibility parameters that facilitate a more precise estimation of the required sample size, specifically within the distinct population of tracheostomized individuals requiring lung reexpansion therapy.

Statistical Analysis: All analyses will be conducted using an intention-to-treat analysis, taking into account the treatment received by each patient in each group following randomization. If a patient's health condition changes and they require invasive ventilatory support for more than 24 consecutive hours or are unable to participate in the intervention, they will be excluded based on exclusion criteria. Blinding will be lifted, and such cases will not be included in the analysis.

For data presentation, for variables with a normal distribution, the measure of central tendency summarizing the data will be the mean, and the standard deviation will be used as a measure of dispersion. When the distribution is non-normal, data will be summarized using the median and interquartile range for continuous variables. Categorical variables will be reported as percentages and presented in frequency tables.

Continuous variables will be analyzed using a Student's t-test for normally distributed data or the Mann-Whitney test for non-parametric data. Categorical variables will be compared using the chi-square test or Fisher's exact test.

To test secondary hypotheses 1 and 2, which state that the use of PED in addition to conventional management is a safe and effective strategy for improving postoperative oxygenation and lung volumes in tracheostomized patients, a comparison between the PED intervention and conventional management alone will be conducted for patients requiring lung reexpansion. This comparison will be achieved using repeated measures analysis of variance (ANOVA) or the non-parametric Friedman test, as appropriate.

For oxygenation, variables such as oxygen saturation (SaO2), arterial oxygen pressure (PaO2), and the ratio of arterial oxygen pressure to inspired oxygen fraction (PaFiO2) measured in arterial gases will be used. For lung volumes, measurements will include inspiratory vital capacity (IVC), IVC with PED, and tidal volume (Vt) as measured by the spirometer. Pulmonary pressures will involve maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP). These measurements, taken at different postoperative time points, will be compared using repeated measures analysis of variance (ANOVA) or the non-parametric Friedman test, as appropriate.

Regarding secondary hypothesis 3, the proportion of patients with postoperative pulmonary complications between the comparison groups from intervention to the end of follow-up will be analyzed using the chi-square test or Fisher's exact test, as needed, to establish statistical significance.

A significance level of p<0.05 will be considered statistically significant. All analyses will be conducted using STATA version 15.7.10.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older.
* Patients with a tracheostomy tube equipped with a functional cuff.
* Patients exhibiting spontaneous breathing for a period exceeding 24 hours.
* Patients requiring lung reexpansion techniques (Postoperative period following thoracic or high abdominal surgery, thoracic trauma, rib fracture, among others).
* Chest imaging confirming the absence of pulmonary parenchyma alterations.

Exclusion Criteria:

* Presence of signs of respiratory distress.
* Alteration in consciousness and loss of decision-making autonomy.
* Cervical spinal cord injury up to T1.
* Muscular weakness due to neuro-demyelinating or peripheral nerve disease.
* Complete dependence on ventilatory support.
* Intracranial pressure greater than 20 mmHg.
* Poorly controlled pain with a Visual Analog Scale (VAS) score of 5 or more.
* Presence of nausea or vomiting.
* Active hemoptysis.
* Pulmonary edema.
* Decompensated congestive heart failure New York Heart Association (NYHA) III-IV.
* Severe physical deconditioning.
* Chronic Obstructive Pulmonary Disease (COPD) Gold E.
* Patients for whom lung reexpansion techniques are contraindicated (pulmonary bullae, pulmonary fistulas, unresolved pneumothorax or hemothorax, medically managed primary spontaneous pneumothorax, platelet count <50,000, among others).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Lung volumes | At three different time points: Day one, day three and day six following the removal of invasive ventilatory support
  Describe the lung volumes through measurements with a Wright respirometer in tracheostomized patients requiring lung reexpansion therapy, where the use of PED plus conventional management is compared to conventional management alone.

SECONDARY OUTCOMES:
Arterial oxygen pressure | At three different time points: Day one, day three and day six following the removal of invasive ventilatory support
  Describe oxygenation through arterial blood sample in tracheostomized patients requiring lung reexpansion therapy, where the use of PED plus conventional management is compared to conventional management alone
Postoperative pulmonary complication | Follow-up throughout hospitalization and up to 28 days from randomization
  Describe the frequency/proportion of postoperative pulmonary complications in tracheostomized patients requiring lung reexpansion therapy, where the use of PED plus conventional management is compared to conventional management alone

CONTACTS AND LOCATIONS:
Overall Officials: MAURICIO VELASQUEZ GALVIS, Study Chair — Fundacion Clinica Valle del Lili

IPD SHARING:
Plan to Share IPD: No
The Clinical Research Center (CRC) of the Fundacion Valle del Lili will generate and maintain all records related to patient selection, inclusion, and data tracking for the study.